CLINICAL TRIAL: NCT02357433
Title: Reduccion de la Mortalidad Mediante Plasma-Adsorción en Shock séptico (ROMPA)
Brief Title: Mortality Reduction in Septic Shock by Plasma Adsorption
Acronym: ROMPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Circumstances beyond the course of the trial have produced a change in the conditions of recruitment unacceptable to the ROMPA researchers
Sponsor: Francisco Colomina Climent (Other)
Responsible Party: Sponsor-Investigator, Francisco Colomina Climent, MD, Hospital Universitario San Juan de Alicante
Organization: Hospital Universitario San Juan de Alicante (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 01-2015_R
Record Dates: First submitted 2015-01-23; First posted 2015-02-06 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

ARMS (2):
- High doses CPFA (Experimental): High doses CPFA (coupled plasma-filtration adsorption) with AMPLYA™ (BELLCO ITALY): >0.20 L/kg/day of plasma treated in the first 3 days after randomization
  Interventions: Device: High Doses CPFA
- Control Group (No Intervention): Standard practice

INTERVENTIONS:
Device: High Doses CPFA
  Arms: High doses CPFA

SUMMARY:
The study objective is to clarify whether the application of high doses CPFA (Coupled Plasma-Filtration Adsorption) in addition to the current clinical practice is able to reduce hospital mortality in septic shock patients in intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the ICU in septic shock
* all patients that develop septic shock while in the ICU

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Estimated life expectancy (due to comorbidities) less than 90 days
* Presence of relative or absolute contraindications to CPFA
* Absence of informed consen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | 28 days

SECONDARY OUTCOMES:
time resolution of septic shock | within the first 28 days
  normalization of lactate, and the decrease in vasoactive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Colomina, MD, Principal Investigator — Hospital Universitario de San Juan de Alicante
Locations (10):
- Spain (10):
  - Hospital de Vinalopó, Elche, Alicante
  - Hospital de la Vega Baja, Orihuela, Alicante
  - Hospital Universitario de San Juan de Alicante, Sant Joan d'Alacant, Alicante
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital de la Plana, Villarreal, Castellon
  - Hospital General Universitario de Santa Lucia, Cartagena, Murcia
  - Hospital Frances De Borja de Gandia, Gandia, Valencia
  - Hospital Lluis Alcanyis, Xátiva, Valencia
  - Hospital General Universitario de Alicante, Alicante

REFERENCES:
- [Derived] Gimenez-Esparza C, Portillo-Requena C, Colomina-Climent F, Allegue-Gallego JM, Galindo-Martinez M, Molla-Jimenez C, Anton-Pascual JL, Marmol-Peis E, Dolera-Moreno C, Rodriguez-Serra M, Martin-Ruiz JL, Fernandez-Arroyo PJ, Blasco-Ciscar EM, Canovas-Robles J, Gonzalez-Hernandez E, Sanchez-Moran F, Solera-Suarez M, Torres-Tortajada J, Palazon-Bru A, Gil-Guillen VF. The premature closure of ROMPA clinical trial: mortality reduction in septic shock by plasma adsorption. BMJ Open. 2019 Dec 3;9(12):e030139. doi: 10.1136/bmjopen-2019-030139. PMID 31796477
- [Derived] Colomina-Climent F, Gimenez-Esparza C, Portillo-Requena C, Allegue-Gallego JM, Galindo-Martinez M, Molla-Jimenez C, Anton-Pascual JL, Rodriguez-Serra M, Martin-Ruiz JL, Fernandez-Arroyo PJ, Blasco-Ciscar EM, Canovas-Robles J, Herrera-Murillo M, Gonzalez-Hernandez E, Sanchez-Moran F, Solera-Suarez M, Torres-Tortajada J, Nunez-Martinez JM, Martin-Langerwerf D, Herrero-Gutierrez E, Sebastian-Munoz I, Palazon-Bru A, Gil-Guillen VF. Mortality Reduction in Septic Shock by Plasma Adsorption (ROMPA): a protocol for a randomised clinical trial. BMJ Open. 2016 Jul 12;6(7):e011856. doi: 10.1136/bmjopen-2016-011856. PMID 27406647